CLINICAL TRIAL: NCT00316485
Title: Diagnosis, Evaluation and Treatment of Patients in Need of Third Molar Removal
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060144; 06-D-0144
Record Dates: First submitted 2006-04-19; First posted 2006-04-20 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-01-28

CONDITIONS: Wisdom Teeth
Keywords: Bone; Microbiology; Dental Pulp Stem Cell; Wisdom Teeth; Biopsy; Third Molar Extraction

SUMMARY:
Under this study, patients who require removal of their third molars (wisdom teeth) will be diagnosed, evaluated and treated. In addition, tooth, bone and gum tissue samples will be collected for use in bone, wound healing, microbiology and genetic research.

Patients 16-50 years of age who require wisdom tooth removal may be eligible for this study. Participants may have one or all of their wisdom teeth removed at one time. The surgery is done under local anesthetic. In addition, conscious sedation may be administered, if the patient wishes.

Besides wisdom tooth removal, patients are asked to donate a small sample of jaw bone (from the lining of the inner wall of the tooth socket) and gum tissue (from the area of the surgical site). The samples are collected at the same time as the tooth extraction. The bone sample is about the size of a pencil point (1.5 millimeters wide and 3 millimeters long) and the gum tissue sample is 1 millimeter. Removal of these samples should not cause any additional discomfort or increase the time required for the surgery or for healing.

DETAILED DESCRIPTION:
OBJECTIVE:

The objective of this protocol is to obtain oral tissue for analysis by various research groups at the National Institutes of Health (NIH).

STUDY POPULATION:

The protocol will enroll a convenience sample of 1,000 subjects between the ages of 18 to 50 years who are in need of third molar (wisdom tooth) extraction.

STUDY DESIGN:

Subjects will report to the National Institutes of Dental and Craniofacial Research (NIDCR) for up to three visits. The first study visit will involve a screening evaluation to determine protocol eligibility. Eligible subjects will be invited back for a second visit for wisdom tooth extraction and collection of oral tissue for research purposes. All subjects will remain on the protocol for three weeks after surgery, and they will have the option to schedule a follow-up visit to the NIH for post-operative evaluation.

OUTCOME MEASURES:

This study does not involve any outcome measurements.

ELIGIBILITY:
* INCLUSION CRITERIA

<TAB>

1. Males and females aged 18 to 50 years
2. Evidence of need for third molar extraction as determined by medical and dental history, as well as clinical and radiographic evaluation
3. Willing to provide at least one wisdom tooth for research purposes
4. Willing to provide one or more of the following tissue types for research purposes:

   Excessive gingival tissue around extraction sockets

   Oral tissues from the floor of the mouth, cheek, palate and/or lateral border of the tongue

   Small biopsies of alveolar bone from the sockets that surround the wisdom teeth
5. America Society of Anesthesiologists (ASA) status I or II

EXCLUSION CRITERIA

1. Pregnant or nursing
2. Clinical signs of infection and/or inflammation, or acute pain at any extraction site at the time of the screening evaluation
3. Known bleeding disorders or conditions associated with bleeding, including Hemophilia, von Willebrand disease, protein C/S deficiency, antithrombin III deficiency, and liver disease.
4. Currently using anticoagulation (blood thinning) medications, including but not limited to warfarin (Coumadin), ticlopidine (Ticlid) and clopidogril (Plavix). Subjects who are currently taking Aspirin and non-steroidal anti-inflammatory drugs (NSAIDs) may be eligible for enrollment.
5. Known or suspected allergy or adverse reaction to any of the agents used for local anesthesia, suture material, or conscious sedation medications
6. Surgical removal of the wisdom teeth is expected to be unusually difficult based on panoramic radiograph. Indicators of unusual difficulty include increased depth of tooth impaction, extreme angulation of a tooth, and close proximity of a tooth to the inferior alveolar nerve canal and/or maxillary sinus.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 718 (Actual)
Dates: Start 2006-04-14; Study Completion 2013-01-28

CONTACTS AND LOCATIONS:
Overall Officials: Carol W Bassim, D.M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Foster JS, Palmer RJ Jr, Kolenbrander PE. Human oral cavity as a model for the study of genome-genome interactions. Biol Bull. 2003 Apr;204(2):200-4. doi: 10.2307/1543559. PMID 12700154
- [Background] Palmer RJ Jr, Gordon SM, Cisar JO, Kolenbrander PE. Coaggregation-mediated interactions of streptococci and actinomyces detected in initial human dental plaque. J Bacteriol. 2003 Jun;185(11):3400-9. doi: 10.1128/JB.185.11.3400-3409.2003. PMID 12754239
- [Background] Kolenbrander PE, Egland PG, Diaz PI, Palmer RJ Jr. Genome-genome interactions: bacterial communities in initial dental plaque. Trends Microbiol. 2005 Jan;13(1):11-5. doi: 10.1016/j.tim.2004.11.005. PMID 15639626